CLINICAL TRIAL: NCT06052917
Title: Impact Study of the Decision Aid DECIdE on the Decisional Conflict of Primary Care Patients About Optional Prescription Drugs.
Brief Title: DECIdE, Shared DECIsion in hEalth : the Real-life Impact Study
Acronym: DECIdE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RESP-IR 2021 VAILLANT-ROUSSEL; 2022-A00071-42 (Other: 2022-A00071-42)
Record Dates: First submitted 2023-09-13; First posted 2023-09-25 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Decision Making, Shared
Keywords: primary care; decision aid; decisional conflict
MeSH Terms: interventions — Health

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with waiting list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DECIdE (Experimental): General practitionners and pharmacists will propose to their patients, complaining of a common symptom for which a drug is usually prescribed or dispensed, to discuss this drug and the symptom in order to reach a shared decision, using DECIdE as a support, on whether to take it or choose another alternative.
  Interventions: Other: DECIdE
- routine without decision aid (No Intervention): General practitionners and pharmacists will prescribe or dispense to their patients, complaining of a common symptom, the drug they usually use and advise them or discuss the benefits and risks as they are used to doing.

INTERVENTIONS:
Other: DECIdE — DECIdE is a decision aid. Its a communication tool to help health providers as general practitioners or community pharmacists, to practice shared medical decision about optional prescription drug. DECIdE provide robust scientific data about benefit and risks associated to the drug under consideration. DECIdE was built based on the consensus of potentials users ( care providers and patients ), tested on users testing and finally validated by a expert consensus ( DELPHI method).
  Other Names: Shared DECIsion in hEalth
  Arms: DECIdE

SUMMARY:
The aim of the DECIdE study is to evaluate the effect of a decision aid (the DECIdE tool) for shared decision making concerning optional prescription drugs on the level of uncertainty-certainty or comfort-inconfort (= decisional conflict) experienced by patients, compared with a condition of routine care without the use of a decision aid.

General practitionners and pharmacists will propose to their patients, complaining of a common symptom for which a drug is usually prescribed or dispensed, to discuss this drug and the symptom in order to reach a shared decision on whether to take it or choose another alternative.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 consulting a general practitioner or community pharmacy
* Patient complaining of a symptom or requesting a optional prescription drug (clinical situations and medicines pre-defined by expert consensus)
* First use of DECIdE with the healthcare professional for this situation
* Agreeing to take part in the study and to sign the written consent form
* Speaks and understands French

Exclusion Criteria:

* minor patients
* Patients under guardianship, curatorship or safeguard of justice
* Pregnant or breast-feeding women
* Second use of the DECIdE tool in the same situation / for the same drug
* Refusal to take part in the study
* Patient not affiliated to a medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
decisional conflict | Day 1
  decisional conflict scale score

SECONDARY OUTCOMES:
effect on decisional conflict categories | day 1
  decision conflict scale scores for each category
effect on health professionals' decisional conflict | day 1
  health professionals' decision conflict scale
effect on the final choose drug | day 1
  Rate of change in patient choice of therapeutic option after use of the tool
medical and economic impact of the choice of drug | day 1
  price of the chosen option
Identify for which type of patient DECIdE reduces decisional conflict | day 1
  age, sex, socio economic category of patient for which the decisional conflict scale is the more reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Vaillant-Roussel, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU Clermont-ferrand, Clermont-Ferrand
  - Département de Médecine Générale, UFR Médecine, Université Grenoble Alpes, Grenoble
  - Collège des Universités de Médecine Générale de Lyon, faculté de médecine Lyon Est, Lyon
  - Département de Médecine Générale de St-Etienne, Faculté de Médecine Jacques Lisfranc, Université Jean Monnet, Saint-Etienne